CLINICAL TRIAL: NCT04810247
Title: Pilot Trial to Enhance Intervention Effects on Weight and Shape Concern Among Women With Higher Body Weight
Brief Title: Targeting Body Image Among Women of Higher Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kayloni Olson, Assistant Professor (Research), The Miriam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K23DK124578 (NIH)
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Results first posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Obesity; Overweight; Body Image
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Body Project intervention (Experimental)
  Interventions: Behavioral: Body Project

INTERVENTIONS:
Behavioral: Body Project — The Body project is a dissonance based intervention designed to target negative body image among adolescent females. The intervention is delivered in small groups of 5-10 individuals over 4, one-hour group sessions. This program will be iteratively revised for use among adult women with weight/shape concern and higher body weight.

SUMMARY:
The goal of this study is to modify the evidence-based Body Project intervention to more powerfully target weight and shape concern among women with BMI between 25-40 using exploratory sequential mixed methodology (using both quantitative and focus group data). Initial modifications to the intervention will be made to incorporate content targeting weight stigma and to ensure the materials are developmentally appropriate for adult women. Then a small group (n=5-10) of women with high weight and shape concern will receive the 4 week body project intervention; we will collect pre-post questionnaire data on weight and shape concern, thin ideal and weight stigma, and use ecological momentary assessment to examine in-the-moment thoughts about weight and shape. The body project intervention will then be revised using this information in combination with participant feedback elicited during a focus group session. The next iteration of the intervention will then be tested in another small group of n=5-10; it is estimated that it will take 4-6 iterations to achieve a more robust intervention program that is acceptable to the target sample. Subgroups (race/ethnicity, BMI class) will be evaluated to ensure suitability across groups.

DETAILED DESCRIPTION:
Women with overweight or obesity, over the age of 25, who report high weight and shape concern and a desire to lose weight will be recruited from the community. Participants will be recruited and enrolled in cohorts of 5-10 individuals, with a focus on ensuring that each group has approximately 50% women of color (i.e., identify as non-white).

Participants will attend, with all individuals in their cohort, the four weekly body project intervention sessions led by a trained facilitator. Each session is approximately 60 minutes long and relies on guided discussion and group activities to engage participants. In between group meetings, participants will be given exercises to complete prior to the next session. The intervention content will be modified prior to the first cohort in order to identify factors relevant for body image among women who would medically benefit from weight loss (e.g., internalized weight bias). The active ingredients will remain the same while modifying content and assignments or exercises to enhance effects among the target population.

Participants will complete a baseline assessment of self-report surveys and a 7-day ecological momentary assessment period. All assessment procedures must be complete prior to the first group meeting. After the fourth and final group meeting, participants will complete a second assessment including self-report surveys and a 7-day EMA period. The data collected from the pre and post-assessments will be used to shape the focus group script. Within four weeks of the last group meeting, participants will attend a focus group meeting led by a facilitator who was not involved in intervention delivery to better understand the participant experience with the intervention content. Key changes may include expanding content to address contextual factors that cause negative weight/shape-related thoughts among women with overweight or obesity and to target weight stigma (internalized), modifying exercises that were reviewed negatively, and incorporating explicit discussion of weight management.

Following the focus group, the intervention will be revised using the quantitative and qualitative data collected from each cohort. The process will be repeated to refine the intervention through iterative testing with small groups of individuals (n≤10). It is anticipated that approximately 4-6 groups will be required. Upon completion of all study procedures, participants will receive information and resources for healthy weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Female
* BMI between 25-40
* EDE-Q weight concern subscale>4
* EDE-Q shape concern subscale>4.25
* Personal use of cell phone
* Able to engage in moderate intensity activity
* Desire for weight loss

Exclusion Criteria:

* No eating disorder history
* Not pregnant
* Not breastfeeding
* No delivery within 9 months
* No substance abuse disorder
* No weight loss medication or history of bariatric surgery
* No other weight loss program participation

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The current study is limited to individuals who identify as female.
Enrollment: 46 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Body Project Intervention: The Body project is an evidence-based intervention designed to target negative body image among adolescent females. This program will be iteratively revised.
  Body Project: The Body project is a dissonance based intervention designed to target negative body image among adolescent females. The intervention is delivered in small groups of 5-10 individuals over 4, one-hour group sessions. This program will be iteratively revised.
Period: Overall Study
Arm/Group | Body Project Intervention
Started | 46
Completed | 39
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Body Project Intervention
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 24
  More than one race | 5
  Unknown or Not Reported | 0
EDE-Q Shape concern subscale [Mean (Standard Deviation); unit: units on a scale] — The Shape concern subscale of the EDE-Q is comprised of the average of 8-items with possible scores ranging from 0-6. Higher scores reflect greater shape concern.
  units on a scale | 5.21 (0.64)
EDE-Q weight concern subscale [Mean (Standard Deviation); unit: units on a scale] — The weight concern subscale of the EDE-Q is comprised of the average of 5-items with possible scores ranging from 0-6. Higher scores reflect greater weight concern.
  units on a scale | 4.59 (0.76)
Internalized weight bias [Mean (Standard Deviation); unit: units on a scale] — Internalized weight bias is calculated by taking the average value of the 10-item Weight Bias Internalization Scale (this excludes item 1 consistent with standards in the field). Possible scores range from 1-7 with higher scores reflecting greater internalized weight bias.
  units on a scale | 5.41 (1.1)
Internalized thin ideal [Mean (Standard Deviation); unit: units on a scale] — Internalized thin ideal is a subscale of the SATAQ-4. It is calculated by taking the average of 5 subscale items and scores can range from 1-5. Higher scores reflect greater internalized thin ideal.
  units on a scale | 3.45 (0.83)

OUTCOME MEASURES:

1. Primary Outcome: EDE-Q Weight and Shape Concern
Description: Participants were eligible for the study if they reported a shape concern score greater than or equal to 4.25 and a weight concern score greater than or equal to 4.0. Clinically significant change in weight and shape concern was defined as no longer meeting study eligibility on just one subscale or on both subscale (shape concern score <4.25; weight concern score <4.0). This outcome reports the number of participants who met this clinical milestone and no longer met criteria for enrollment.
Time Frame: 4 weeks
Population: Completers
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6: The Body Project intervention was iteratively revised between each cohort.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 9 | 7 | 0 | 8 | 7 | 8
Participants
  No longer meet enrollment criteria on the weight subscale or on the shape subscale | 3 | 6 | 0 | 3 | 4 | 5
  No longer meet enrollment criteria for either the shape subscale OR the weight subscale | 2 | 1 | 0 | 2 | 1 | 0

2. Primary Outcome: Sociocultural Attitudes Towards Appearance Questionnaire-4
Description: Internalized thin ideal is a subscale of the SATAQ-4. Scores can range from 1-5. Higher scores reflect greater internalized thin ideal
Time Frame: Baseline and 4 weeks
Population: Only completers analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 9 | 7 | 0 | 8 | 7 | 8
score on a scale
  Baseline | 3.98 (0.67) | 3.2 (0.86) |  | 3.2 (0.96) | 3.26 (0.75) | 3.6 (1.06)
  4 week | 3.8 (0.85) | 2.77 (0.96) |  | 2.85 (0.66) | 2.86 (1.06) | 3.55 (0.69)

3. Primary Outcome: Weight Bias Internalization Scale
Description: Internalized weight bias is calculated by taking the average value of the 10-item Weight Bias Internalization Scale (this excludes item 1 consistent with standards in the field). Possible scores range from 1-7. Higher scores reflect greater internalized weight bias.
Time Frame: Baseline and 4 weeks
Population: Only completers included in analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 9 | 7 | 0 | 8 | 7 | 8
score on a scale
  Baseline | 5.84 (0.87) | 5.09 (1.23) |  | 5.6 (0.76) | 5.0 (1.38) | 5.53 (1.13)
  4 weeks | 5.37 (1.11) | 4.06 (1.39) |  | 4.75 (1.39) | 4.21 (1.24) | 4.56 (1.00)

4. Secondary Outcome: Momentary Weight and Shape Concern
Description: Participants rated how negative their thoughts were about weight and shape since the previous prompt (on a 0-10 scale) 6 times per day for 7 days at baseline and following treatment. Individual participant responses were presented graphically and coded as representing a general decrease, increase, or no change in negative weight/shape-related thoughts from baseline to 4 weeks.
Time Frame: Baseline and four weeks
Population: Only completers
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 9 | 7 | 0 | 8 | 7 | 8
Participants
  Decreased weight/shape-related negative thoughts | 6 | 5 |  | 7 | 6 | 6
  No change in weight/shape-related negative thoughts | 3 | 2 |  | 0 | 1 | 1
  Increased weight/shape-related negative thoughts | 0 | 0 |  | 1 | 0 | 1

5. Secondary Outcome: Qualitative Feedback
Description: Attendance at focus group. Following the four-week modified Body Project intervention, participants were asked to attend a meeting to provide feedback on their experience in the intervention.
Time Frame: within 4 weeks of intervention completion
Population: Only completers
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 9 | 7 | 0 | 8 | 7 | 8
Participants | 8 | 6 |  | 4 | 5 | 3

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Body Project Intervention
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/46

LIMITATIONS AND CAVEATS:
Cohort 3 was discontinued by the PI due to low engagement. After the first group meeting, only 1 of 5 enrolled individuals was engaged/actively participating. Delivering the intervention one-on-one is not consistent with protocol and the group environment is conceptually an active ingredient of the intervention (and an important component per Focus Group feedback). Therefore, the study team decided to discontinue all study procedures for this group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-31): https://cdn.clinicaltrials.gov/large-docs/47/NCT04810247/Prot_SAP_000.pdf